CLINICAL TRIAL: NCT06595849
Title: Acceptability, Feasibility, and Effectiveness of a Four-Week Feeling Tone Mindfulness Course
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1005240113_Study2
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mindfulness; Depression; Anxiety; Stress; Wellbeing; Self-compassion
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This is a single-arm trial, where all participants will be assigned to the intervention group.
  Interventions: Behavioral: 4-week feeling tone intervention program

INTERVENTIONS:
Behavioral: 4-week feeling tone intervention program — Participants will take part in a 4-week mindfulness of feeling tone intervention program taught by a registered mindfulness teacher, who is also a registered clinical psychologist. The intervention program includes 4 sessions, with each session lasting for about 2 hours. The program is taught in Cantonese, in a group setting, live online (via Zoom). Participants will practice meditation practices during the session, explore themes of the week, review and explore their meditation experiences. They will also practice meditation practices daily for at least 30 minutes at home, with meditation audio recordings provided by the teacher.

SUMMARY:
This is an academic research study aiming to explore the acceptability, feasibility, and effectiveness of a four-week feeling tone mindfulness course on equanimity, mindfulness, self-compassion, and mental health outcomes.

DETAILED DESCRIPTION:
The four-week feeling tone mindfulness course is an adapted version of a mindfulness intervention program recently developed by Professor Mark Williams and colleagues. This study aims to explore the acceptability, feasibility, and effectiveness of a four-week feeling tone mindfulness course on equanimity, mindfulness, self-compassion, and mental health outcomes (e.g., depression, anxiety, stress, wellbeing) in a Hong Kong population.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above
* speak and understand Cantonese as well as written Chinese to a level where the participant can fully take part in the course without the need for translation support
* have means to access online teleconferencing meeting software (e.g., Zoom), online surveys, online intervention materials, and Short Message Service (SMS) or WhatsApp messenger

Exclusion Criteria:

* moderately severe or severe depressive or anxiety symptoms
* diagnosed with bipolar disorder or bipolar affective disorder (type I or type II) or ever experienced a manic/hypomanic episode
* diagnosed with schizophrenia/ psychosis or ever experienced a psychotic episode
* diagnosed with dementia/ neurocognitive disorders/ neurological disorders
* diagnosed with intellectual disability
* diagnosed with other neurodevelopmental disorders
* experience of a traumatic event that is currently affecting the potential participants
* recent bereavement, major loss, or stressful life events
* suicidal
* alcohol or drug abuse
* currently experiencing other mental or physical health condition, or life condition that might affect potential participants' participation in the course
* prior experience of taking part in the feeling tone intervention as a course participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mindfulness (Five Facet Mindfulness Questionnaire - 20) | 4-week; 8-week
  The 20-item Five Facet Mindfulness Questionnaire - 20 (FFMQ-20) will be used to measure mindfulness. Possible score range is 20 to 100, where higher scores indicate higher mindfulness.
Equanimity (Equanimity Scale) | 4-week; 8-week
  The 16-item Equanimity Scale (ES-16) will be used to measure equanimity. Possible score range is 16 to 80, where higher scores indicate higher equanimity.
Self-compassion (Sussex-Oxford Compassion for the Self Scale) | 4-week; 8-week
  The 20-item Sussex-Oxford Compassion for the Self Scale (SOCS-S) will be used to measure self-compassion. Possible score range is 20 to 100, where higher scores indicate higher self-compassion.

SECONDARY OUTCOMES:
Depression (Patient Health Questionnaire - 9) | 4-week; 8-week
  The nine-item Patient Health Questionnaire - 9 (PHQ-9) will be used to measure depression. Possible score range is 0 to 27, where higher scores mean more severe depression.
Anxiety (Generalized Anxiety Disorder - 7) | 4-week; 8-week
  The seven-item Generalized Anxiety Disorder-7 (GAD-7) will be used to measure anxiety. Possible score range is 0 to 21, where higher scores indicate more severe anxiety.
Stress (Perceived Stress Scale - 10) | 4-week; 8-week
  The 10-item Perceived Stress Scale - 10 (PSS) will be used to measure stress. Possible score range is 0 to 40, where higher scores indicate higher perceived stress.
Wellbeing (Short Warwick-Edinburgh Mental Wellbeing Scale) | 4-week; 8-week
  The seven-item Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) will be used to measure wellbeing. Possible score range is 0 to 35, where higher scores mean higher mental wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Hoi Chun Lok, MSocSc(CP), Principal Investigator — Department of Psychology, The University of Hong Kong
Locations (1):
- Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong